CLINICAL TRIAL: NCT05663892
Title: Drug-drug Interaction Study Between Bictegravir/Emtricitabine/Tenofovir Alafenamide and Feminizing Hormones in Trans Women Living With HIV
Brief Title: Drug-Drug Interaction Study in Trans Women Living With HIV
Acronym: T-DDI
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Maple Leaf Research (Other)
Responsible Party: Principal Investigator, Mona Loutfy, Dr., Maple Leaf Research
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CTN 331
Record Dates: First submitted 2022-11-27; First posted 2022-12-23 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Hiv; Transgenderism
Keywords: HIV; Feminizing Hormone Therapy; Transgender Women; Antiretroviral Therapy; Drug-Drug Interaction
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Transsexualism | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Investigational Population (Group 1) - Trans women living with HIV (Experimental): Trans women living with HIV, taking:
  * Biktarvy
  * Oral 17(Beta)-Estradiol
  Interventions: Drug: Biktarvy 50/200/25 Tab; Drug: Estradiol Tablets
- Comparator Population (Group 2) - Cis Women Living with HIV (Active Comparator): Cis women living with HIV, taking:
  -Biktarvy
  Interventions: Drug: Biktarvy 50/200/25 Tab
- Comparator Population (Group 3) - Trans Women Living without HIV (Active Comparator): Trans women living without HIV, taking:
  -Oral 17(Beta)-Estradiol
  Interventions: Drug: Estradiol Tablets

INTERVENTIONS:
Drug: Biktarvy 50/200/25 Tab — As the HIV ART, the combination of B/F/TAF, known as Biktarvy®, which is a widely available Single Tablet Regimen (STR) approved by Health Canada is the drug under investigation. Participants in groups 1 and 2 will either have to already be taking B/F/TAF or will be required to switch to it at baseline and they will self-administer B/F/TAF once daily in the morning, with or without food. Participants taking their dosage at night will be required to switch to a morning dose at the screening visit.
  Arms: Comparator Population (Group 2) - Cis Women Living with HIV; Investigational Population (Group 1) - Trans women living with HIV
Drug: Estradiol Tablets — Oral 17(beta)-estradiol as the estrogen and an anti-androgen (pharmaceutical [e.g., spironolactone, cyproterone, finasteride, leuprolide, bicalutamide, dutasteride] and/or surgical [orchiectomy] and/or medical [hypogonadism]).Doses of estradiol range from 1 mg to a maximum of 6 mg per day.
  Participants must take 2 mg until the Month 2 Visit. Trans women participants in both groups 1 and 3 must divide their dose to twice a day (BID) if they are taking > 2 mg per day and take 2 mg in the morning and the rest of the dosing in the evening. Participants who are only taking 2mg of estradiol once daily at night must switch their dosing to the morning. Participants who either crush or take the oral estradiol sublingually must switch to swallowing the tablet orally from the day after the screening visit until the Month 2 visit, otherwise the estradiol concentrations will be markedly higher.
  Other Names: Oral 17(beta)-estradiol
  Arms: Comparator Population (Group 3) - Trans Women Living without HIV; Investigational Population (Group 1) - Trans women living with HIV

SUMMARY:
Introduction: Transgender (trans) women have been found to be at higher risk of and to be disproportionally affected by HIV. Trans women with HIV have also been found to have low usage and adherence rates to antiretroviral therapy (ART). Both healthcare providers and trans women, themselves, have expressed concerns of drug-drug interactions (DDIs) between ART drugs and feminizing hormones, which have in turn been shown to contribute to low rates of ART usage amongst trans women with HIV. The objective of this DDI study is to investigate the pharmacokinetic effects of the common feminizing hormone regimens (oral estradiol with an anti-androgen (pharmaceutical and/or surgical and/or medical) on the antiretroviral combination bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) and vice versa.

Methods and Analysis: Participants will be assigned to three groups: group 1 will include 15 trans women with HIV who are taking feminizing hormones and ART (investigational group); group 2 will include 15 premenopausal cis women with HIV taking ART (ART control group); group 3 will include 15 trans women without HIV taking feminizing hormones (hormone control group). Women with HIV will have to be virally suppressed for at least three months and they will have to already be taking B/F/TAF or have their current ART regimen switched to B/F/TAF at baseline. Trans women participants will be required to be on 2 mg oral estradiol or higher and an anti-androgen (pharmaceutical, medical or surgical). Plasma ART drug concentrations will be sampled at the 2-month visit and compared among trans women with HIV on feminizing hormones and premenopausal cis women with HIV. Serum estradiol and total testosterone concentrations will be sampled at the baseline and month 2 visits and compared among trans women with and without HIV. If successful, this trial will serve to provide empirical evidence regarding a lack of, or presence of DDIs between B/F/TAF and feminizing hormones.

Dissemination: The findings will be disseminated through publication in peer-reviewed journals as well as presented at national and international conferences and community groups.

DETAILED DESCRIPTION:
Introduction: Transgender (trans) women have been found to be at higher risk of and to be disproportionally affected by HIV for multiple biologic and social reasons. Trans women living with HIV have also been found to have low usage and adherence rates to antiretroviral therapy (ART). Both healthcare providers and trans women, themselves, have expressed concerns of drug-drug interactions (DDIs) between ART drugs and feminizing hormones, which have in turn been shown to contribute to low rates of ART usage amongst trans women living with HIV. The objective of this DDI study is to investigate the pharmacokinetic effects of the common feminizing hormone regimens (oral estradiol with an anti-androgen (pharmaceutical and/or surgical and/or medical)) on the antiretroviral combination bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) and vice versa.

Methods and analysis: Participants will be assigned to three groups: group 1 will include 15 trans women living with HIV who are taking feminizing hormones and ART (investigational group); group 2 will include 15 premenopausal cis women living with HIV taking ART (ART control group); group 3 will include 15 trans women living without HIV taking feminizing hormones (hormone control group). Women living with HIV will have to be virally suppressed for at least three months and they will have to already be taking B/F/TAF or have their current ART regimen switched to B/F/TAF at baseline. Trans women participants will be required to be on 2 mg oral estradiol or higher and an anti-androgen (pharmaceutical, medical or surgical). Plasma ART drug concentrations will be sampled at the 2-month visit and compared among trans women living with HIV on feminizing hormones and premenopausal cis women living with HIV. Serum estradiol and total testosterone concentrations will be sampled at the baseline and month 2 visits and compared among trans women living with and without HIV. The primary endpoints are B/F/TAF pharmacokinetic parameters (Cmin, Cmax and AUC) between trans and cis women living with HIV at month 2 and the estradiol concentrations (Cmin, C4h, Cmax and AUC) and the proportions of the month 2 C4h that are within target (200 to 735 pmol/L) between trans women living with and without HIV at month 2. Other endpoints will include the mean estradiol and testosterone concentrations at baseline and the difference between baseline and month 2 estradiol pre-dose and C4h, satisfaction with feminizing hormones, HIV viral load, adherence, adverse events, patient-reported outcomes (i.e., symptoms), satisfaction with ART regimen and health status. If successful, this trial will serve to provide empirical evidence regarding a lack of, or presence of DDIs between B/F/TAF and feminizing hormones.

Dissemination: The findings will be disseminated through publication in peer-reviewed journals as well as presented at national and international conferences and community groups.

ELIGIBILITY:
Investigational Population (Group 1) - Trans Women Living with HIV

Inclusion Criteria

1. Is a trans woman or person with transfeminine experience (individual assigned male sex at birth who currently identifies as a woman or person with transfeminine experience and is at any stage of medical, social, or legal transition);
2. Is 18 years of age or older;
3. Is living with HIV;
4. Is currently taking combination ART and has been taking these medications for at least 3 months prior to the screening visit;
5. Is willing to adjust their ART dosing to the morning if they are currently taking it at night for at least 28 days before the baseline visit until the completion of the Month 2 visit;
6. Has had an undetectable viral load for at least 3 months on at least two occasions, where most recent (within 12 months including screening) VL<40 copies/mL and second (within 24 months) VL<200 copies/mL with no suggestion of relevant ART drug resistance prior to screening;
7. Is willing to switch to or stay on B/F/TAF for the duration of the study (i.e., 6 months);
8. Is currently taking oral estradiol (2 mg or higher) and an anti-androgen (pharmaceutical [e.g., spironolactone, cyproterone, finasteride, leuprolide, bicalutamide, dutasteride] and/or surgical [orchiectomy] and/or medical [hypogonadism]) and has been taking these medications together at the current dose for at least 3 months prior to the screening visit; AND:

   1. Is willing to adjust their oral estradiol dosing to twice a day if they are taking > 2 mg per day (which is currently recommended as best practice) for at least 28 days before the baseline visit until the completion of the Month 2 visit, with the morning dose set at 2 mg (remaining dose can be taken at night), OR;
   2. If their estradiol dosing is 2 mg per day and they are currently taking their estradiol at night, they must be willing to switch their dosing to the morning for at least 28 days before the baseline visit until the completion of the Month 2 visit;
   3. Is willing to swallow their oral estradiol if they are currently taking it sublingually or crushing it for at least 28 days before the baseline visit and until the completion of the Month 2 visit;
   4. Is willing to keep their anti-androgen (if applicable) medication(s) unchanged until the completion of the Month2 visit;
9. If taking progesterone, is willing to keep the same medication/dose until the completion of the Month 2 visit and must have been taking that dose for at least 3 months prior to the screening visit;
10. Is willing and able to provide full consent for their participation.

Exclusion Criteria

1. Is clinically unable to switch ART to B/F/TAF based on their physician's opinion;
2. Is taking hormonal non-prescription or natural health products in addition to feminizing hormone therapy;
3. Has significant underlying diseases which could worsen due to their participation, or affect their ability to follow the study procedures;
4. Has kidney or liver impairment (ALT > 5X normal; serum creatinine [eGFR] < 30 mL per minute);
5. Is taking medications known to interact with feminizing hormones, B/F/TAF, or its individual components or has taken such medications within the past 28 days prior to baseline (List of prohibited medications in Appendix B1).
6. Has a known hypersensitivity to bictegravir (BIC), emtricitabine (FTC), tenofovir alafenamide (TAF) or to any ingredient in the formulation.

Comparator Population (Group 2) - Cis Women Living With HIV Inclusion Criteria

1. Is a cis woman (individual assigned female sex at birth who currently identifies as a woman);
2. Is of reproductive age and 18 years of age or older;
3. Is living with HIV;
4. Has a regular period (every 24 - 35 days), or if period is irregular or absent, it is due to the administration of a progesterone only hormone contraceptive (see Appendix B1); or if uterus removed (hysterectomy), ovarie(s) remain functional (FSH level<27.0 IU/L);
5. Is currently taking combination ART and has been taking these medications for at least 3 months prior to screening;
6. Is willing to adjust their ART dosing to the morning if they are currently taking it at night for at least 28 days before the baseline visit until the completion of the Month 2 visit;
7. Has had an undetectable viral load for at least 3 months on at least two occasions, where most recent (within 12 months including screening) VL<40 copies/mL and second (within 24 months) VL<200 copies/mL with no suggestion of relevant ART drug resistance prior to screening;
8. Is willing to switch to or stay on B/F/TAF for the duration of the study (i.e., 6 months);
9. Is willing and able to provide full consent for their participation.

Exclusion Criteria

1. Is clinically unable to switch B/F/TAF based on their physician's opinion;
2. Is pregnant or is planning on getting pregnant for the duration of the study;
3. Has undergone surgery to remove their ovaries (i.e. oophorectomy) or has a condition in which their ovaries produce little or no estrogen (i.e. primary ovarian insufficiency, hypogonadism) or does not have ovaries naturally (i.e. unilateral ovarian absence); total hysterectomy is allowed as long as ovaries are intact and functional;
4. Is taking an estrogen containing or conjugated estrogens hormonal therapies; IUD and progesterone only contraception are allowed (See Appendix B1/2 for list for both prohibited and allowed contraceptives);
5. Has significant underlying diseases which could worsen due to their participation, or affect their ability to follow the study procedures;
6. Has kidney or liver impairment (ALT > 5X normal; serum creatinine [eGFR] < 30 mL per minute);
7. Has a known hypersensitivity to bictegravir (BIC), emtricitabine (FTC), tenofovir alafenamide (TAF) or to any ingredient in the formulation.
8. Is taking medications known to interact with B/F/TAF, or its individual components or has taken such medications within the past 28 days prior to baseline (List of prohibited medications in Appendix B1/2).

Comparator Population (Group 3) - Trans Women Living Without HIV Inclusion Criteria

1. Is a trans woman or person with transfeminine experience (defined as individual assigned male sex at birth who currently identifies as a woman or person with transfeminine experience irrespective of medical, social, or legal transition);
2. Is 18 years of age or older;
3. Is HIV negative at screening;
4. Is currently taking oral estradiol (2mg or higher) and an anti-androgen (pharmaceutical [i.e., spironolactone, cyproterone, finasteride, leuprolide, bicalutamide, dutasteride] and/or surgical [orchiectomy] and/or medical [hypogonadism]) and has been taking these medications at the current dose for at least 3 months prior to the screening visit, AND:

   1. Is willing to adjust their oral estradiol dosing to twice a day if they are taking > 2 mg per day (which is currently recommended as best practice) for at least 28 days before the baseline visit until the completion of the Month 2 visit, with the morning dose set at 2 mg (remaining dose can be taken at night) OR;
   2. If their estradiol dosing is 2 mg per day and they are currently taking their estradiol at night, they must be willing to switch their dosing to the morning for at least 28 days before the baseline visit until the completion of the Month 2 visit;
   3. Is willing to swallow their oral estradiol if they are currently taking it sublingually or crushing it for at least 28 days before the baseline visit until the completion of the Month 2 visit;
   4. Is willing to keep their anti-androgen (if applicable) medication(s) unchanged until the completion of the Month2 visit;
5. If taking progesterone, is willing to keep their dose the same until the Month 2 visit and must have been taking that dose for at least 3 months prior to the screening visit;
6. Is willing and able to provide full consent for their participation.

Exclusion Criteria

1. Is taking hormonal non-prescription or natural health products in addition to feminizing hormone therapy;
2. Has taken HIV pre-exposure prophylaxis (PrEP) (i.e, TDF/FTC or TAF/FTC) or HIV post-exposure prophylaxis (PEP) in the prior 28 days from baseline and plans to continue during the study;
3. Has significant underlying diseases which could worsen due to their participation, or affect their ability to follow the study procedures;
4. Has kidney or liver impairment (ALT > 5X normal; serum creatinine [eGFR] < 30 mL per minute);
5. Is taking medications known to interact with feminizing hormones or has taken such medications within the past 28 days prior to baseline (List of prohibited medications in Appendix B1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is open to:
  * Transgender women or persons with transfeminine experience, taking feminizing hormone therapy (oral estradiol)
  * Cisgender women.
Enrollment: 45 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
BIC, FTC, and TAF minimum plasma concentrations. | Month 2
  Minimum plasma concentrations (Cmin) of BIC, FTC, and TAF concentrations will be compared between trans women living with HIV (group 1) and premenopausal cis women living with HIV (group 2).
BIC, FTC, and TAF maximum plasma concentrations. | Month 2
  Maximum plasma concentrations (Cmax) of BIC, FTC, and TAF concentrations will be compared between trans women living with HIV (group 1) and premenopausal cis women living with HIV (group 2).
BIC, FTC, and TAF area under the curve (AUC) plasma concentrations. | Month 2
  AUC plasma concentrations of BIC, FTC, and TAF will be compared between trans women living with HIV (group 1) and premenopausal cis women living with HIV (group 2).
2h PBMC and DBS TFV-DP and FTC-TP concentrations. | Month 2
  PBMC and DBS TFV-DP and FTC-TP concentrations done at 2h after ingestion of medications will be compared between trans women living with HIV (group 1) and premenopausal cis women living with HIV (group 2).
Minimum serum concentrations (Cmin) of estradiol. | Month 2
  Estradiol Cmin at month 2 will be compared between groups 1 and 3.
4 hour serum concentration (C4h) of estradiol | Month 2
  Estradiol C4h at month 2 and the proportions of the month 2 C4h that are within target (200 to 735 pmol/L) and will be compared between groups 1 and 3.
Maximum serum concentrations (Cmax) of estradiol | Month 2
  Estradiol Cmax at month 2 will be compared between groups 1 and 3.
Estradiol serum concentration area under the curve (AUC) | Month 2
  Estradiol AUC at month 2 will be compared between groups 1 and 3.

SECONDARY OUTCOMES:
Baseline estradiol pre-dose serum concentration (Cmin) and comparison to month 2 | Months 0 & 2
  Baseline estradiol pre-dose concentrations, and these will be compared between groups 1 and 3 and assessed to see the proportion that meets target. The baseline estradiol pre-dose concentrations will be taken on variable ART regimens for the trans women living with HIV; the month 2 estradiol pre-dose concentrations will be taken from the trans women living with HIV who are taking B/F/TAF; and the change in estradiol pre-dose concentrations from baseline to month 2 in those who switched to B/F/TAF will be compared to those who did not and to those in group 3.
Baseline estradiol C4h serum concentration and comparison to month 2 | Months 0 & 2
  Baseline estradiol C4h concentrations, and these will be compared between groups 1 and 3 and assessed to see the proportion that meets target. The baseline estradiol C4h concentrations will be taken on variable ART regimens for the trans women living with HIV; the month 2 estradiol C4h concentrations will be taken from the trans women living with HIV who are taking B/F/TAF; and the change in estradiol C4h concentrations from baseline to month 2 in those who switched to B/F/TAF will be compared to those who did not and to those in group 3.
Baseline total testosterone serum concentration and comparison to month 2 | Months 0 & 2
  Baseline total testosterone concentrations, and these will be compared between groups 1 and 3 and assessed to see the proportion that meets target. The baseline total testosterone concentrations will be taken on variable ART regimens for the trans women living with HIV; the month 2 total testosterone concentrations will be taken from the trans women living with HIV who are taking B/F/TAF; and the change in total testosterone concentrations from baseline to month 2 in those who switched to B/F/TAF will be compared to those who did not and to those in group 3.
FEM-SQ questionnaire score | Months 0, 2 & 6
  Total score on the Feminizing Medical Gender Affirmation Satisfaction Scale (FEM-SQ), a questionnaire for measuring satisfaction with medical gender affirmation, will be compared between groups 1 and 3 throughout the study period. The FEM-SQ is a new questionnaire developed by our team through mixed-methods survey development including expert consultation and focus groups with 23 trans women (version 1), semi-structured interviews with over 10 trans women (version 2), and quantitative data collection (survey administration) with 300 trans women (version 3). For the importance sub-scale the minimum score is 0 and the maximum score is 85. For the satisfaction sub-scale the minimum score is 18 and the maximum sub score is 90 with higher scores meaning the participant is satisfied with their feminizing hormone therapy.
Proportion of patient with an undetectable HIV-RNA. | Months 0, 2 & 6
  Proportion of patients with an undetectable HIV-RNA (<40 copies/mL) will be compared between groups 1 and 2 throughout the study period.
ART adherence using theMedication Adherence Self-Reported Inventory (MASRI) | Months 0, 1, 2 & 6
  ART adherence will be assessed at each visit for groups 1 and 2 using a validated visual analogue scale (VAS) of ART use, the MASRI, over the prior month at each visit. The instructions for the VAS read: 'put a cross on the line below at the point showing your best guess about how much medication you have taken in the last month. We would be surprised if this was 100% for most people, e.g., 0% means you have taken no medication; 50% means you have taken half your medication; 100% means you have taken every single dose of medication'. The VAS ranges from 0 to 100% in 10% intervals.
Frequency of BIC, FTC, and TAF related adverse events | Months 1, 2 & 6
  Frequency and severity of B/F/TAF related adverse effect for participants in groups 1 and 2 who have changed to B/F/TAF at each follow-up visit.
  Adverse effects will be recorded using the NIAID standardized toxicity grading system (Appendix D) and will be reported as a frequency and proportion of with any adverse effect, any grade 2 or higher and any requiring stopping the treatment.
Patient reported outcomes (PROs) using the HIV Symptom Index Distress Module (HSIDM) | Months 0, 1, 2 & 6
  PROs will be assessed for groups 1 and 2 at all study visits using the HSIDM at baseline, months 2 and 6. However, since the scale does not mention HIV and asks about symptoms solely, group 3 participants will be asked to complete it at baseline and month 2. Participants are asked about their experience with each of 20 symptoms during the past 4 weeks using a 5-point, Likert-type scale; therefore the minimum score is 0 and and maximum is 100. A higher score would mean that the participant has had a lot of symptoms and it has bothered them a lot.
Satisfaction with ART Regimens using the HIVTSQ | Months 0, 2 & 6
  We will be asking about satisfaction with ART regimen using the HIV Treatment Satisfaction Questionnaire (HIVTSQ). There are two versions of the HIVTSQ that have been developed. At the baseline, month 2 and month 6 visits, the 10-item HIVTSQ status version (HIVTSQs) will be used. The HIVTSQc will be used in addition to the HIVTSQs at month 6. The questionnaires are both scored out of 66, the HIVTSQs has a range from 0 to 66 with a higher score meaning that one is more satisfied with their treatment. Item number 12 is not included in the composite score, it is stand alone. The HIVTSQc ranges from -33 to +33.
Participant health status using the SF-36 | Months 0, 2 & 6
  Participant health status in all groups will be assessed using the SF-36 at baseline and month 2, which allows us to convert to a utility and conduct cost-effectiveness analyses in the future, if desired. The SF-36 will be repeated for Groups 1 and 2 at the 6-month visit. The SF-36 consists of eight scale scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health). These eight scale scores are the weighted sums of the questions in their section and then each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. SF-36 is interpreted in ascending fashion with lower scores equating to more disability and higher scores meaning less disability. The individual scale scores and overall scale score are most often reported as a mean and standard deviation (SD).

OTHER OUTCOMES:
Basic sociodemographic variables | Month 0
  Basic sociodemographic variables will be collected such as age [to be reported as a median with interquartile range (IQR)] and race/ethnicity [White, African, Caribbean Black (ACB), Indigenous or Other (N/%)].
Clinical variables | Months 0 & 2
  Clinical variables will include weight (median/IQR), height (median/IQR), body mass index (median/IQR), and hepatitis B or C infection (N/%).
FHT regimens | Month 0
  For the trans women participants, dose of estradiol will be recorded (N/% and median/IQR), which anti-androgen/orchiectomy/medical is used (N/%) and its dose (N/%), and whether gender affirming surgery has taken place, more specifically orchiectomy which can impact testosterone concentrations.
HIV clinical history | Month 0
  For participants living with HIV, duration of HIV infection (median/IQR), duration of ART (median/IQR), which ART regimen they are currently taking, baseline VL (median/IQR), baseline CD4 count (median/IQR) will be collected.
Menstrual history | Month 0, 2 & 6
  For cis women, a menstrual history will be recorded including if their cycles are regular (N/%).

CONTACTS AND LOCATIONS:
Overall Officials: Mona Loutfy, MD, MPH, Principal Investigator — Maple Leaf Research
Locations (1):
- Maple Leaf Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT05663892/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT05663892/ICF_001.pdf